CLINICAL TRIAL: NCT04365595
Title: Recovery in Patients With SARS-CoV-2 Associated Respiratory Failure
Brief Title: SARS-CoV-2 Associated Respiratory Failure Recovery (COVID-19 CAir)
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-00745
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: SARS-CoV 2; COVID
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SARS-CoV-2 associated respiratory failure: Participants will receive a daily HrQoL questionnaire on their personal smartphone using the docdok health application during 3 months. A selection of participants will furthermore receive a custom-built home disease monitoring device during 1 month. Both procedures start at least 4 weeks after hospital discharge.
  Interventions: Other: Questionnaires, spirometry

INTERVENTIONS:
Other: Questionnaires, spirometry — Questionnaires targeting health-related quality-of-life, symptoms, anxiety and depression

SUMMARY:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is the cause of the current pandemic of coronavirus disease (COVID-19) that can lead to respiratory failure requiring oxygen therapy. Some patients develop acute respiratory distress syndrome (ARDS) and may die despite intensive care therapy. Currently it is unknown a) how fast patients recover after being discharged from hospital and b) what underlying predictors may influence recovery.

DETAILED DESCRIPTION:
Study aims:

* To evaluate subjective and objective recovery after discharge from hospital in patients with respiratory failure due to COVID-19.
* To identify risk factors for COVID-19 associated respiratory failure and prolonged recovery

ELIGIBILITY:
Inclusion Criteria:

* hospitalization at University Hospital Zurich due to COVID-19 infection
* hospital discharge max. 4 weeks ago
* requiring supplemental oxygen

Exclusion Criteria:

* <18 years
* non-German speaking
* no smartphone access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with SARS-CoV-2 associated respiratory failure
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2021-02-17 (Actual)

PRIMARY OUTCOMES:
Health-related quality-of-life | 3 months
  European Quality of Life - 5 Dimensions - 5 Levels Instrument (EQ-5D-5L). Scoring: Index ranges from 1 to <0, with lower scores indicating more limitations.

SECONDARY OUTCOMES:
Anxiety and depression | 3 months
  Hospital Axiety and Depression Score (HADS). Scoring: Scores range from 0 to 42, with higher scores indicating more anxiety or depression symptoms.
Symptom burden | 3 months
  COPD Assessment Test (CAT). Scoring: Scores range from 0-40, with higher scores indicating more symptoms due to respiratory limitations.
Spirometry | 1 month
  Forced expiratory volume in one second (FEV1) in liters and percent predicted.
Spirometry | 1 month
  Forced vital capacity (FVC) in liters and percent predicted.

CONTACTS AND LOCATIONS:
Overall Officials: Christian F Clarenbach, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
on reasonable request

REFERENCES:
- [Derived] Kohlbrenner D, Kuhn M, Stussi-Helbling M, Nordmann Y, Spielmanns M, Clarenbach CF. Longitudinal Smartphone-Based Post-hospitalisation Symptom Monitoring in SARS-CoV-2 Associated Respiratory Failure: A Multi-Centre Observational Study. Front Rehabil Sci. 2021 Nov 24;2:777396. doi: 10.3389/fresc.2021.777396. eCollection 2021. PMID 36188784